CLINICAL TRIAL: NCT02514499
Title: Multiplex Testing for Evaluation of Breast Cancer Risk, Longitudinal Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Screening
Other Study IDs: UPCC 07914
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: BRCA1/2 Negative
Keywords: patients
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Questionnaires

SUMMARY:
The overall goal of the proposed research is to evaluate the uptake of testing and longitudinal risks and benefits of multiplex testing for cancer susceptibility in BRCA1/2 negative patients. This model will inform the selection of the outcomes and potential mediators and moderators of these outcomes, to inform the debate over utility, risks, and benefits of clinical incorporation of multiplex testing for breast cancer susceptibility.

ELIGIBILITY:
Inclusion Criteria:

* 1. Women and men (at least 18 YO) 2. English speaking AND 3. Negative for BRCA1 and BRCA2 mutations

Exclusion Criteria:

1. Non English speaking patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350
Dates: Start 2014-07; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Completion of questionnaires | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States